CLINICAL TRIAL: NCT07346586
Title: Effect of an Individualized Urinary Catheter Management Strategy on the Safety and Efficacy of Early Catheter Removal After Mid-Low Rectal Cancer Surgery: A Single-Center Randomized Controlled Trial
Brief Title: Effect of Individualized Catheter Management on Early Removal After Rectal Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yuchen Guo, Ph.D., Prof., The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICCAUT-3
Record Dates: First submitted 2025-12-21; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urinary Catheters; Rectal Cancer; Urinary Retention
Keywords: Urinary Retention; Rectal Cancer; Catheter
MeSH Terms: conditions — Rectal Neoplasms; Urinary Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized Management Group (Experimental): Participants assessed by the AUR risk prediction model immediately postoperatively. High-risk patients receive prophylactic tamsulosin until catheter removal. All patients have their catheter removed at 4:00 AM on postoperative day 1.
  Interventions: Behavioral: Individualized Management Group
- 24-Hour Removal Group (Experimental): Participants do not receive prophylactic tamsulosin. The urinary catheter is removed uniformly at 4:00 AM on postoperative day 1.
  Interventions: Behavioral: 24-Hour Removal Group
- 48-Hour Removal Group (Active Comparator): Participants do not receive prophylactic tamsulosin. The urinary catheter is removed uniformly at 4:00 AM on postoperative day 2.
  Interventions: Behavioral: 48-Hour Removal Group

INTERVENTIONS:
Behavioral: Individualized Management Group — Participants assessed by the AUR risk prediction model immediately postoperatively. High-risk patients receive prophylactic tamsulosin until catheter removal. All patients have their catheter removed at 4:00 AM on postoperative day 1.
  Arms: Individualized Management Group
Behavioral: 24-Hour Removal Group — Participants do not receive prophylactic tamsulosin. The urinary catheter is removed uniformly at 4:00 AM on postoperative day 1.
  Arms: 24-Hour Removal Group
Behavioral: 48-Hour Removal Group — Participants do not receive prophylactic tamsulosin. The urinary catheter is removed uniformly at 4:00 AM on postoperative day 2.
  Arms: 48-Hour Removal Group

SUMMARY:
This study aims to systematically evaluate the safety and efficacy of different early urinary catheter removal strategies following radical resection of mid-low rectal cancer. Current clinical practice faces controversy regarding the optimal timing of catheter removal (24 hours vs. 48 hours) and lacks precise preventive measures for patients at high risk of postoperative acute urinary retention (AUR). To address these issues, this study is designed as a three-arm randomized controlled trial, directly comparing three management protocols: catheter removal at 24 hours postoperatively, catheter removal at 48 hours postoperatively, and an individualized strategy guided by a predictive model (i.e., preventive administration of tamsulosin to high-risk AUR patients prior to catheter removal). The primary endpoint is the rate of recatheterization within 7 days after the initial removal, with secondary endpoints comprehensively assessing urinary tract infections, voiding function, and postoperative complications. The ultimate goal is to provide high-quality evidence-based medical evidence to establish a precise and standardized clinical pathway for individualized postoperative catheter management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a preoperative pathological confirmation of rectal malignant tumor.
2. Preoperative colorectal CT or rectal MRI confirming that the lower edge of the tumor is located in the rectum within 10 cm from the anal verge (including rectal and anal canal lesions).
3. Patients scheduled to undergo laparoscopic or robot-assisted radical total mesorectal excision (TME).

Exclusion Criteria:

1. History of previous abdominal surgery involving the rectum/sigmoid colon/left colon, bladder resection or partial resection, prostate surgery (in males), or hysterectomy (in females).
2. History of urethral trauma, intracranial surgery, spinal surgery, cerebral infarction with limb dysfunction, or Parkinson's disease.
3. Inability to void urethrally preoperatively due to any reason (e.g., ureteral puncture, ureterostomy).
4. Previously diagnosed overactive bladder syndrome, prior AUR or voiding dysfunction, or diabetic cystopathy.
5. Preoperative assessment indicating potential need for combined resection of other pelvic organs during surgery, including the bladder, prostate, uterus and cervix, or vagina (excluding simple adnexectomy in females).
6. Preoperative assessment indicating potential need for lateral pelvic lymph node dissection.
7. Preoperative renal insufficiency (serum creatinine level >133 μmol/L).
8. Patients undergoing emergency surgery.
9. Male patients with preoperative benign prostatic hyperplasia requiring medication.
10. Presence of indwelling ureteral stents, ureteral stenosis, or bilateral hydronephrosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1545 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2029-11-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of recatheterization within 7 days after the initial catheter removal | Rate of recatheterization within 7 days after the initial catheter removal
  Recatheterization will be performed if the patient meets any of the following criteria for acute urinary retention (AUR) after catheter removal:
  Criterion 1: Inability to void spontaneously within 6 hours of catheter removal, with a post-void residual volume (PVR) >300ml on bladder ultrasound, which persists (>300ml) after a trial of oral tamsulosin and an additional 4-hour observation period.
  Criterion 2: Persistent and strong urge to void with minimal urine output, frequency, sensation of bladder fullness, bladder pain, or new-onset incontinence, coupled with a PVR >300ml on bladder ultrasound.
  Criterion 3: Patient request for recatheterization due to severe discomfort from bladder distension, provided that the volume of urine immediately obtained exceeds 200ml.

SECONDARY OUTCOMES:
Incidence of Catheter-Associated Urinary Tract Infection (CAUTI). | within 1 days after the initial catheter removal
  Catheter-Associated Urinary Track Infection is defined as the inflammatory response of the urinary tract epithelium to bacterial invasion related to catheter placement. The diagnosis must simultaneously satisfy the following two criteria: 1) Urinalysis indicates that the urinary bacterial count exceeds the upper limit of the normal range, and 2) Urine culture is positive.
  Incidence of Catheter-Associated Urinary Tract Infection (CAUTI) is calculated as a ratio: UTI cases occurring after first catheter removal divided by the total number of enrolled participants.
Time to First Successful Voiding after Catheter Removal | within 1 days after the initial catheter removal
  The time to first void after catheter removal is defined as the period from the time of catheter removal to the time when the patient voids spontaneously, measured in hours.
Voiding function assessed by the ICIQ-SF questionnaires after catheter removal | within 2 days after the initial catheter removal
  ICIQ-SF(International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form), minimum / maximum (total score ) is 0 to 21, higher scores means worse outcome(greater severity/impairment from urinary incontinence).
Voiding function assessed by the lPSS questionnaires after catheter removal | within 2 days after the initial catheter removal
  IPSS(International Prostate Symptom Score) , Minimum / maximum (symptom score): 0 to 35 the single quality-of-life question is scored 0 to 6 ("delighted" → "terrible"), where higher means worse QoL; higher scores in total indicates worse outcome (more severe urinary symptoms); Mild (IPSS 0-7): Symptom severity is considered mild, and active treatment is usually not required unless the patient is bothered by symptoms.Moderate (IPSS 8-19): Symptoms are moderate; treatment options (e.g., medication, minimally invasive therapy) should be discussed based on the patient's condition and preferences. Severe (IPSS 20-35): Symptoms are severe and typically require active intervention (e.g., medication, surgery) to improve quality of life.
Incidence, types, and severity (graded by Clavien-Dindo classification) of postoperative complications within 30 days. | within 30 days postoperatively
  The Clavien-Dindo classification includes, but is not limited to, intra-abdominal hemorrhage, gastrointestinal bleeding, anastomotic leakage, chyle leakage, surgical site infection (intra-abdominal infection and incisional infection), intestinal obstruction, postoperative diarrhea, pulmonary infection, urinary tract infection, cardiovascular accident, cerebrovascular accident, and thrombotic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After we complete our study
Access Criteria: Researchers may provide legitimate justification and supporting documentation.